CLINICAL TRIAL: NCT04781582
Title: Comparison of Lung Volume Reduction Surgery Versus Bronchoscopic Lung Volume Reduction in Patients With Homogenous Emphysema: A Prospective Randomized Trial
Brief Title: LVRS Versus BLVR in Patients With Homogenous Emphysema, CLUB-HE Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Clemens Aigner, Professor of Thoracic Surgery, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-9518-BO
Record Dates: First submitted 2021-02-25; First posted 2021-03-04 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Emphysema or COPD
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive | interventions — Pneumonectomy

STUDY DESIGN:
Intervention Model Description: single center, 1:1 randomized, open label, controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lung volume reduction surgery arm (Active Comparator): Bilateral videothoracoscopic lung volume reduction surgery by wedge resection. Unilateral procedures are possible in case of severe adhesions or intraoperative instability. In these cases a staged approach with contralateral LVRS within 3 months is possible.
  Interventions: Procedure: Lung volume reduction surgery
- Bronchoscopic lung volume reduction arm (Active Comparator): Primarily unilateral bronchoscopic lung volume reduction by endobronchial valves. If a bilateral procedure is feasible it must be performed within 3 months after the first intervention.
  Interventions: Procedure: Bronchoscopic lung volume reduction

INTERVENTIONS:
Procedure: Lung volume reduction surgery — Surgical lung volume reduction
  Arms: Lung volume reduction surgery arm
Procedure: Bronchoscopic lung volume reduction — Bronchoscopic lung volume reduction by endobronchial valves
  Arms: Bronchoscopic lung volume reduction arm

SUMMARY:
This is a prospective randomized clinical trial comparing surgical and bronchoscopic lung volume reduction in patients with advanced homogeneous emphysema suitable for both procedures.

DETAILED DESCRIPTION:
Lung volume reduction surgery (LVRS) as well as bronchoscopic lung volume reduction (BLVR) provide functional improvements in selected patients with homogenous emphysema and pronounced hyperinflation. A direct comparison of LVRS and BLVR in patients with homogenous emphysema is not available, thus the study will provide important data to guide treatment selection in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* COPD III-IV
* Age ≥ 18 years
* FEV1 < 50% predicted after bronchodilatation
* Significant hyperinflation (TLC >100% predicted, RV > 200% predicted, RV/TLC > 60%)
* Non-smoker or ex-smoker for > 3 months (documented by cotinine testing)
* 6 MWT >150 m and ≤ 450m
* MRC dyspnea score > 3
* Homogenous emphysema as assessed by HR-CT (< 15% difference in emphysema destruction score between target lobe and ipsilateral lobe) [16, 17]
* Uni- or bilateral collateral ventilation (CV) negative result assessed fissure completeness>95% in QCT and confirmed by a bronchoscopic procedure (Chartis©)
* Optimal medical therapy for > 3months, sufficient rehabilitation status with no need for further training/rehabilitation or rehabilitation within 6 months prior to intervention.
* Body Mass Index (BMI) > 18, but < 35 kg/m2
* Daily dose of prednisone ≤ 10mg

Exclusion Criteria:

* Contraindication against either LVRS or BLVR and/or to surgery and bronchoscopy in general
* Major comorbidities limiting survival
* Age ≥ 80 years
* Nicotine abuse within 3 months (documented by cotinine testing)
* Predominance of either left or right lung of >70% in perfusion SPECT scintigraphy
* FEV1 and/or DLCO <20% predicted (post bronchodilatation)
* Untreated Hypoxemia (PaO2 < 50 mmHg)
* Untreated Hypercapnia (PaCO2 > 50 mmHg)
* Significant pulmonary fibrosis or bronchiectasis
* Destroyed/vanished lung on HR-CT
* Previous chest surgery or bronchoscopic interventions
* Pulmonary hypertension (sPAP > 35 mmHg)
* Active waiting list for lung transplantation
* Patient is not able to understand and willing to sign a written informed consent document.
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2021-06-08 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Change in FEV1 compared to baseline (deltaFEV1) | 6 months post intervention
  Percent change in FEV1

SECONDARY OUTCOMES:
Change in BODE Index (Body mass index, airflow obstruction, dyspnoea and exercise capacity in chronic obstructive pulmonary disease) | 3, 6 months post intervention
  Combined score including BMI, FEV1, 6 MWT, MRC dyspnoea score; range 0 (best) - 10 (worst)
Change in TLC | 3, 6 months post intervention
  Percent change in Total Lung Capacity
Change in RV | 3, 6 months post intervention
  Percent change in Residual Volume
Change in RV/TLC | 3, 6 months post intervention
  Percent change in RV/TLC ratio
Change in DLCO | 3, 6 months post intervention
  Percent change in diffusion capacity
Change in systolic pulmonary artery pressure | 6 months post intervention
  measured by echocardiography
Changes in health-related quality of life measured by SGRQ | 3, 6 months post intervention
  St. George´s Respiratory Questionnaire (score 0-100, higher scores indicating more limitations)
Changes in respiratory health status measured by CAT | 3, 6 months post intervention
  COPD Assessment Test (CAT)
Mortality | 30 days post intervention
  Number of deaths 30 days post intervention
Overall survival | 6 months post intervention
  Percent of patients alive 6 months post intervention
Incidence of (serious) adverse events | Periprocedural, 1, 3, 6 months post intervention
  Number of events periprocedural, 1, 3 and 6 months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Clemens Aigner, Prof. MD, Principal Investigator — Universität Duisburg-Essen
Locations (1):
- University Medicine Essen, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No